CLINICAL TRIAL: NCT03292705
Title: Applying a Person-Centered Approach to Enhance Cognitive Training in Senior Living Community Residents With Mild Cognitive Impairment
Acronym: CogT-PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Vankee Lin, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21AG054810 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Mild Cognitive Impairment
Keywords: cognitive training; person-centered approach
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: A single-blinded, multi-site (4 SLCs) randomized controlled trial of PEP+CCI, vs. control + CCI is involved. For PEP+CCI group, PEP will be implemented for the first 4 weeks, and CCI for the following 6 weeks. For the control + CCI group, an inert control condition, consisting of nothing outside of the ordinary, will be implemented for the first 4 weeks, and CCI for 6 more weeks. Assessments will be conducted by our research team. Separate staff blind to group assignment will conduct post-training and follow-up assessments. All intervention and assessments will occur in private rooms in relevant SLCs.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to the group assignment. The participants will be informed to avoid discussing their intervention activities at the post-training and follow up assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP+CCI (Experimental): PEP: The PEP system is built on a picture-based touch-screen interface on tablet computers. PEP allows users to explore and participate in entertainment, educational, spiritual, and other recreational activities and content personalized according to their interests and preferences. It provides easy access to the Internet and communication applications, and has hundreds of modules spanning music, travel, trivia, games, and religious and inspirational domains.
  CCI. VSOP training will use five training paradigms (Eye for detail, Peripheral challenge, Visual sweep, Double decision, Target tracker) that practice processing speed and attention.
  Intervention format and fidelity The PEP+CCI group will practice PEP for the first 4 weeks and VSOP for the following 6 weeks.
  Interventions: Behavioral: PEP; Behavioral: CCI
- control+CCI (Active Comparator): For the control + CCI group, an inert control condition, consisting of nothing outside of the ordinary, will be implemented for the first 4 weeks, and CCI for 6 more weeks.
  Interventions: Behavioral: CCI

INTERVENTIONS:
Behavioral: PEP — The PEP system is built on a picture-based touch-screen interface on tablet computers. PEP allows users to explore and participate in entertainment, educational, spiritual, and other recreational activities and content personalized according to their interests and preferences. It provides easy access to the Internet and communication applications, and has hundreds of modules spanning music, travel, trivia, games, and religious and inspirational domains. For instance, if music is among a person's lifelong interests, the system provides access to multiple music genres through jukebox, karaoke and therapeutic music applications that can be tailored to a particular activity and by individual interest (for instance, a preference for classic jazz). As another example, for someone who likes travel or visiting new places, the interface offers access to Google Earth, guided tours, slide shows and regional facts and history.
  Arms: PEP+CCI
Behavioral: CCI — VSOP training will use five training paradigms (Eye for detail, Peripheral challenge, Visual sweep, Double decision, Target tracker) that practice processing speed and attention. All exercises share visual components and focus on accuracy and fast reaction times. Participants respond either by identifying what object they see or where they see it on the screen. The training will automatically adjust the difficulty of each task based on the participant's performance, ensuring that the participants always operate near their optimal capacity. The training programs will automatically record the percentage of completion of each game and scores.

SUMMARY:
Computerized cognitive interventions (CCIs) have been increasingly widely implemented among older adults with mild cognitive impairment (MCI). However, the efficacy of CCIs in maintaining or improving older adults' cognitive and functional health has been modest and highly variable. Older individuals' attitudes toward technology use may help explain some of the variability in CCI effects. The goal of this R21 is to generate proof-of-concept for an intervention that may improve attitudes toward computers among those with MCI, in turn improving engagement with and efficacy of a subsequent CCI. Person-centered care-that is, integrating individuals' preferences throughout the process of intervention--has improved intervention engagement among older persons, including those with MCI. A recent intervention predicated on this person-centered approach is called "personalized engagement program" (PEP). PEP involves a database of individualized computer-led leisure activities. The investigators' recent pilot data in senior living facilities suggest that PEP promotes psychological well-being among older persons with MCI, and may shift computers from dauntingly complex or personally irrelevant devices to familiar, enjoyable technology. These results are consistent with a number of theories indicating that exposure to pleasurable experiences with an object or task improves several dimensions of attitudes, including affective and cognitive components, as well as behavior and motivation. Grounded in both this pilot data and the theory around it, the investigators seek to take the next step in an arc of research ultimately intended to improve the efficacy of CCIs. A small randomized controlled trial (RCT) is proposed to assess whether an initial period of PEP, followed by a standard CCI, improves a) attitudes toward computers, b) engagement with the CCI, and c) cognitive outcomes, compared to an attention control period followed by CCI. Our design involving stratified random assignment of 50 assisted living residents with MCI from 4 senior living facilities to these two groups. The initial phase involves 4 weeks of either attention control or PEP, a "dose" suggested by prior work on attitude change and computers, followed by 6 weeks of CCI for both groups (a period our prior work indicates is sufficient for change in key cognitive domains among this population). This application is the first of which we are aware striving to augment CCIs, which are now ubiquitous, by addressing an attitudinal or affective element of the person, which are often ignored in the cognitive intervention literature. The adjuvant of PEP also answers increasing calls for "personalized" or "person-centered" behavioral interventions with older persons.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ MoCA ≤ 26
* RAVLT Delayed Recall Total Score ≤ 6 (or 1.5 SD below age-corrected norms)
* mild or no active depressive symptoms
* intact or mild deficits in IADL functioning
* if on AD medication (i.e., Memantine or cholinesterase inhibitors), antidepressant, or anxiolytics, no changes of doses in the 3 months prior to recruitment;
* age ≥60 years
* English-speaking
* adequate visual and hearing acuity for testing
* intact decision making capacity.

Exclusion Criteria:

* current enrollment in another cognitive improvement study;
* uncontrollable major depression: or other psychopathology identified by staff or medical records;
* having active legal guardian (indicating impaired capacity for decision making);
* medical history of AD or other types of dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Attitudes Toward Computers Questionnaire Total score | Baseline, End of Weeks 4, End of Week 10, & Week 23
  change of attitudes towards technology across time points
Useful Field of View | Baseline, End of Week 10, & Week 23
  change of visual speed of processing and attention across time points
Executive Function | Baseline, End of Weeks 4, End of Week 10, & Week 23
  change of executive function across time points
Brief Visuospatial Memory Test | Baseline, End of Weeks 4, End of Week 10, & Week 23
  change of visuospatial memory across time points

SECONDARY OUTCOMES:
Activities of Daily Living-Prevention Instrument | Baseline, End of Weeks 4, End of Week 10, & Week 23
  change of self-perceived functioning in daily living activities across time points
Everyday Problems for Cognitive Challenged Elderly Test | Baseline, End of Weeks 4, End of Week 10, & Week 23
  change of objective functioning in daily living activities across time points

CONTACTS AND LOCATIONS:
Overall Officials: Anne Corriveau, PhD, Study Director — University of Rochester
Locations (2):
- United States (2):
  - Brickstone/Saint John Meadow, Rochester, New York
  - River Edge Manor, Rochester, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin FV, Cottone K, Mcdermott K, Jacobs A, Nelson D, Porsteinsson A, Chapman BP. Attitudes Toward Computers Moderate the Effect of Computerized Cognitive Trainings in Oldest-Old Senior Living Center Residents. Am J Geriatr Psychiatry. 2021 Mar;29(3):285-294. doi: 10.1016/j.jagp.2020.07.001. Epub 2020 Jul 7. PMID 32739240